CLINICAL TRIAL: NCT05426421
Title: Tolerability of Lopinavir Versus Dolutegravir for Children and Adolescents Living With HIV (LoDoCA): a Prospective Cohort Study
Brief Title: Tolerability of Lopinavir Versus Dolutegravir for Children and Adolescents Living With HIV
Acronym: LoDoCA
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); University of Basel (Other); University of Zurich (Other); Baylor International Pediatric AIDS Initiative (Unknown); Lesotho Ministry of Health (Unknown); Baylor College of Medicine Children's Foundation Lesotho (Unknown)
Responsible Party: Sponsor
Other Study IDs: P001-22-1.0; ID37-2022 (Other: National Health Research Ethics Committee (Lesotho)); H-51472 (Other: Institutional Review Board for Baylor College of Medicine and Affiliated Hospitals); 3ZX1422 (Other Grant/Funding Number: University of Basel Research Fund)
Record Dates: First submitted 2022-06-11; First posted 2022-06-22 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: HIV
Keywords: dolutegravir; lopinavir; children; adolescents; paediatric; adverse effects; tolerability; treatment satisfaction; insomnia; sleep; gastrointestinal; depression; human immunodeficiency virus; cohort
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spots
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No actigraphy: Participants will receive viral load testing at transition from LPV/r-based to DTG-based ART, and subsequent routine viral load data will be analysed. Questionnaires will be filled in and dried blood spots collected at transition and at four weeks. Medical history as well as clinical and socio-demographic data will be collected.
- With actigraphy: Participants will receive viral load testing at transition from LPV/r-based to DTG-based ART, and subsequent routine viral load data will be analysed. Baseline actigraphy data will be collected for two weeks prior to transition (actigraphy period 1), and for four weeks after transition (actigraphy period 2 from 0-2 weeks after transition; actigraphy period 3 from 2-4 weeks after transition). Sleep diaries will be filled in during all actigraphy periods. Questionnaires will be filled in and dried blood spots taken at transition as well as two and four weeks after transition. Medical history as well as clinical and socio-demographic data will be collected.

SUMMARY:
Dolutegravir-based antiretroviral therapy is set to be increasingly replace ritonavir-boosted lopinavir-based regimens for the treatment of paediatric HIV. This prospective cohort study aims to compare tolerability, adverse effects, and virological outcomes between the two regimen types using a before-after design. The study is conducted in Lesotho, southern Africa, and includes children and adolescents transitioning from ritonavir-boosted lopinavir-based to dolutegravir-based antiretroviral therapy. It aims to provide detailed information on treatment tolerability and to inform paediatric treatment programmes.

DETAILED DESCRIPTION:
Dolutegravir, an antiretroviral drug to treat HIV, has recently been rolled out on a large scale across much of Africa. With paediatric formulations becoming increasingly available, dolutegravir is set to replace ritonavir-boosted lopinavir as the core agent in paediatric treatment regimens in many countries. While both drugs are well-studied and highly effective, they reportedly differ with regards to their tolerability at least in adults, with ritonavir-boosted lopinavir typically associated with gastrointestinal adverse effects and dolutegravir mostly associated with neuropsychiatric adverse effects including insomnia. Resistance patterns also differ between these two treatment options. However, studies focusing specifically on the tolerability of and adverse effects associated with either drug in children and adolescents are scarce.

This prospective cohort study aims to i) compare treatment satisfaction, health-related quality of life, tolerability, and symptoms or side-effects associated with either drug option, ii) specifically compare sleep outcomes quantified through actigraphy with either drug option, and iii) provide observational evidence on virological outcomes in a resource-limited setting using a before-after design.

The study is conducted at several sites in Lesotho, southern Africa. It enrols children and adolescents <18 years of age who are taking ritonavir-boosted lopinavir-based therapy at enrolment and routinely due to transition to dolutegravir-based therapy as per the national roll-out plan. On the day of transitioning to dolutegravir as well as four weeks thereafter, participants will complete questionnaires on treatment satisfaction, gastrointestinal symptoms, depressive symptoms, and sleep habits. A subset of participants fulfilling additional inclusion criteria will additionally use actigraphy sensors to monitor sleep duration and sleep fragmentation; these individuals will have study visits two weeks before transition to dolutegravir to initiate actigraphy, at transition, as well as two and four weeks after transition, with questionnaires at all but the pre-transition visit and actigraphy (target: at least seven nights with high-quality data) between all visits. For all participants, medical records will be assessed and additional clinical and sociodemographic data collected. A viral load test will be done on the day of transitioning to dolutegravir, and subsequent routine viral load test results (every six months as per national guidelines) will be assessed. Dried blood spots will be taken at all visits, barring the pre-transition visit for those with actigraphy.

This study aims to inform the continued roll-out of dolutegravir replacing ritonavir-boosted lopinavir in paediatric antiretroviral therapy regimens, notably assessing the suitability of a one-size-fits-all approach and providing detailed information on tolerability and adverse effects of either regimen.

ELIGIBILITY:
Inclusion Criteria - general:

* Currently taking ritonavir-boosted lopinavir-containing antiretroviral therapy
* Eligible for dolutegravir-based antiretroviral therapy as per national roll-out/guidelines
* Age < 18 years
* Informed consent (as per consenting procedures)

Exclusion Criteria - general:

* No transition to dolutegravir-based antiretroviral therapy foreseen
* Already enrolled in another study judged as non-compatible by the Principal Investigator or Local Principal Investigator

Inclusion Criteria - actigraphy:

* Enrolled into main cohort
* Age ≥6 and <18 years
* Taking ritonavir-boosted lopinavir-containing antiretroviral therapy for at least 12 weeks
* Last viral load <50 copies/mL and taken within <36 weeks and while taking ritonavir-boosted lopinavir-containing antiretroviral therapy
* Willingness to wear an actimetry sensor every night for at least 7 nights (daytime wearing optional)
* Patient and/or caregiver judged to be able to fulfil requirements (wearing actimetry sensor; filling in sleep diary) by study team member conducting screening
* Stated ability to attend all study visits
* Informed consent (as per consenting procedures)

Exclusion Criteria - actigraphy:

* Intention to transfer out of the study site (and not into a different study site) within 6 weeks
* No actimetry sensor available

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adolescents living with HIV, receiving treatment, and transitioning from ritonavir-boosted lopinavir-based to dolutegravir-based antiretroviral therapy in the context of the national rollout of dolutegravir.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Sleep duration during monitoring period 3 (2-4 weeks post-transition) versus monitoring period 1 (0-2 weeks pre-transition) | [2-4 weeks post-transition] vs [0-2 weeks pre-transition]
  Sleep will be monitored using actigraphy sensors for a subset of participants. There will be three sleep monitoring periods: 0-2 weeks before transition from ritonavir-boosted lopinavir- to dolutegravir-based antiretroviral therapy (period 1), 0-2 weeks after transition, and 2-4 weeks after transition). We will conduct a before-after analysis.
Change in treatment satisfaction, assessed using the HIV Treatment Satisfaction Questionnaire (HIVTSQ) change version (HIVTSQ-c) | 4 weeks post-transition
  10-item scale with each item scored from -3 to +3 (overall range -30 to +30), with higher scores indicating increases in treatment satisfaction

SECONDARY OUTCOMES:
Viral suppression rate among those with virological data | 6 months, 12 months, and 24 months after transition
  Proportion of participants with a viral load <50 copies/mL among all participants with virological data
Engagement in care with viral suppression | 6 months, 12 months, and 24 months after transition
  Proportion of participants with a viral load <50 copies/mL among all participants
Sleep duration during monitoring period 2 (0-2 weeks post-transition) versus monitoring period 1 (0-2 weeks pre-transition) | [0-2 weeks post-transition] vs [0-2 weeks pre-transition]
  Sleep will be monitored using actigraphy sensors for a subset of participants. There will be three sleep monitoring periods: 0-2 weeks before transition from ritonavir-boosted lopinavir- to dolutegravir-based antiretroviral therapy (period 1), 0-2 weeks after transition, and 2-4 weeks after transition). We will conduct a before-after analysis.
Sleep fragmentation | [2-4 weeks post-transition] vs [0-2 weeks pre-transition], and [0-2 weeks post-transition] vs [0-2 weeks pre-transition]
  Sleep will be monitored using actigraphy sensors for a subset of participants. There will be three sleep monitoring periods: 0-2 weeks before transition from ritonavir-boosted lopinavir- to dolutegravir-based antiretroviral therapy (period 1), 0-2 weeks after transition, and 2-4 weeks after transition). We will conduct a before-after analysis.
Treatment satisfaction after vs before transition, assessed using the HIVTSQ status version (HIVTSQ-s) | 4 weeks post-transition vs at transition
  10-item scale with each item scored from 0 to 6 (overall range 0 to 60), with higher scores indicating higher treatment satisfaction. Two time points compared in a before-after analysis.
Gastrointestinal symptoms after vs before transition, assessed using the Gastrointestinal Symptom Rating Scale adapted for protease inhibitors (GSRS-PI) | 4 weeks post-transition vs at transition
  13-item scale with each item scored from 1 to 6, with higher scores indicating greater discomfort. Two time points compared in a before-after analysis.
Depressive symptoms after vs before transition, assessed using the Center for Epidemiological Studies Depression Scale for Children (CES-DC) | 4 weeks post-transition vs at transition
  20-item scale with each item scored from 0 to 3 (overall range 0 to 60), with higher scores indicating higher depressive symptoms. Two time points compared in a before-after analysis.
Sleep outcomes after vs before transition, assessed using the Child Sleep Habits Questionnaire (CSHQ) or Adolescent Sleep Habits Questionnaire (ASHQ) | 4 weeks post-transition vs at transition
  33-item scale (2 items used in two subscales) with each item scored from 1 to 3, with higher scores indicating more sleep problems. Two time points compared in a before-after analysis.
Health-related quality of life after vs before transition, assessed using the KINDL questionnaire | 4 weeks post-transition vs at transition
  24-item scale with each item scored from 1 to five, with higher scores indicating higher health-related quality of life

OTHER OUTCOMES:
Proportion of participants with drug resistance among participants with viraemia while taking dolutegravir | until 24 months after transition
  Classified Stanford HIV drug resistance database (susceptible, potential low-level resistance, low-level resistance, intermediate resistance, high-level resistance) referring to each drug in the current ART regimen
Impact of drug resistance at time of transition on subsequent viral suppression | until 24 months after transition
  Assessment whether resistance at transition predicts subsequent routinely assessed viral load outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brown, PhD, Principal Investigator — University of Basel; Akash Devendra, MBChB, Principal Investigator — Baylor International Paediatric AIDS Initiative
Locations (1):
- Baylor Center of Excellence Maseru, Maseru, Lesotho

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared in a data repository upon publication of results.